CLINICAL TRIAL: NCT02824952
Title: Neo-adjuvant Trial With AZD9291 in EGFRm+ Stage IIIA/B NSCLC - a Phase 2 Open-label Study
Brief Title: Neo-adjuvant Trial With AZD9291 in EGFRm+ Stage IIIA/B NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Nir Peled, Head of Oncology, Shaare Zedek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0432-20-SZMC; 0432-20-SZMC (Other: Shaare Zedek Medical Center)
Record Dates: First submitted 2016-06-29; First posted 2016-07-07 (Estimated); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Lung Cancer, Non-small Cell
Keywords: Tagrisso; AZD9291; EGFRm; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tagrisso 80 mg (Experimental): 80 mg of Tagrisso(AZD9291) will be given every day for 6 or 12 weeks.
  Interventions: Drug: Tagrisso

INTERVENTIONS:
Drug: Tagrisso — taking orally everyday for 6 or 12 weeks.
  Other Names: AZD9291

SUMMARY:
Patients will receive AZD9291 at a dose of 80 mg once daily. Systemic evaluation will be done by PET-CT scan after 6 weeks.

In responding patients AZD9291 will be given orally 80 mg daily for 12 weeks. Non-responding patients will receive AZD9291 for the period of 6 or 12 weeks (according to the results of response assessment at each time-point).

DETAILED DESCRIPTION:
Patients will receive AZD9291 at a dose of 80 mg once daily. Systemic evaluation will be done by PET-CT scan after 6 weeks.

In responding patients AZD9291 will be given orally 80 mg daily for 12 weeks. Non-responding patients will receive AZD9291 for the period of 6 or 12 weeks (according to the results of response assessment at each time-point). All the patients will be followed for 2 years.

The imaging modality used for RECIST v1.1 assessments will be PET-CT scan.

ELIGIBILITY:
Inclusion Criteria.

1. Provision of informed consent prior to any study specific procedures
2. Male or female, aged at least 18 years.
3. Treatment-naïve stage IIIA/B NSCLC with an activating sensitizing EGFR mutation/T790M

   • Uncommon sensitizing EGFR mutations are allowed.
4. Measurable disease by RECIST criteria v1.1.
5. Patients are amenable for curative chemo-radiotherapy.
6. ECOG PS 0/1.

   •total bilirubin less then 1.5 mg/dL, ALT+ AST levels 3 times above the upper normal limit.
7. Normal hematologic, renal and liver function:

   * Absolute neutrophil count over 1500/mm3, platelets over 100,000/mm3, hemoglobin over 9 g/dL;
   * Creatinine concentration less than 1 mg/dL, or creatinine clearance over 60 mL/min;
   * Total bilirubin less than 1.5 mg/dL, ALT and AST levels 3 times above the upper normal limit.
8. FEV-1 more than1 liter.
9. Female patients with reproductive potential must have a negative pregnancy test (serum/urine) prior to starting treatment.
10. All patients with reproductive potential must agree to use barrier contraception methods while receiving the study treatment.

Exclusion criteria

1. EGFR TKI - resistant EGFR mutations (e.g., insertion in exon 20)
2. T790M is allowed.
3. Treatment with any of the following:
4. Prior treatment with any systemic anti-cancer therapy for advanced NSCLC;
5. Prior treatment with an EGFR-TKI;
6. Major surgery within 4 weeks of the first dose of study drug;
7. Treatment with an investigational drug within five half-lives of the compound.
8. Pregnant or lactating women.
9. Inability to sign the informed consent form.
10. Any concurrent and/or other active malignancy that has required systemic treatment within 2 years of first dose of study drug.
11. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses; or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV), uncontrolled diabetes.
12. Inability to swallow the formulated product, malabsorption syndrome, refractory nausea and vomiting that would preclude adequate absorption of AZD9291.
13. Any of the following cardiac criteria:
14. Mean resting corrected QT interval (QTc) >470 msec, obtained from 3 consequent ECGs, using the screening clinic ECG machine-derived QTc value;
15. Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG;
16. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, including unexplained sudden death under 40 years of age in a first-degree relative, or any concomitant medication known to prolong the QTc interval.
17. Any evidence/past medical history of interstitial lung disease (ILD) or radiation pneumonitis which required steroid treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate as defined by RECIST 1.1 | 12 weeks
  assessed by PET-CT

SECONDARY OUTCOMES:
mPFS measured by Kaplan-Meier method. | 2 years
  mPFS measured by Kaplan-Meier method.
Comparing GTV (Gross tumor volume) before and after the neoadjuvant therapy | 2 years
  Comparing GTV (Gross tumor volume) before and after the neoadjuvant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Nir Peled, MD PhD FCCP, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No